CLINICAL TRIAL: NCT02215694
Title: Supplementation of Dual Probiotic Strains, Lactobacillus Curvatus HY7601 and Lactobacillus Plantarum KY1032, Reduced Fasting Triglyceride and Enhanced Apolipoprotein A-V Levels in Nondiabetic and Hypertriglyceridemic Subjects
Brief Title: Supplementation of Dual Probiotic Strains Reduced Fasting Triglyceride and Enhanced Apolipoprotein A-V Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: probiotics_140801
Record Dates: First submitted 2014-08-02; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Hypertriglyceridemia
Keywords: Apolipoprotein A-V; LDL particle size; probiotic; triglyceride
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic group (Experimental): consumed 2g of powder daily containing dual probiotics(Lactobacillus curvatus HY7601 and Lactobacillus plantarum KY1032)
  Interventions: Dietary Supplement: dual probiotics
- placebo group (Placebo Comparator): consumed 2g of powder daily without probiotics
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: dual probiotics — 2g of powder daily containing dual probiotics(Lactobacillus curvatus HY7601 and Lactobacillus plantarum KY1032)
  Other Names: probiotic
  Arms: probiotic group
Dietary Supplement: placebo — 2g of powder daily without probiotics
  Arms: placebo group

SUMMARY:
The purpose of this study is to evaluate the effect of dual probiotic strains containing Lactobacillus curvatus HY7601 and Lactobacillus plantarum KY1032 on triglyceride and apolipoprotein A-V.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study was conducted on 128 nondiabetic and hypertriglyceridemic (Plasma Triglyceride, 150-500 mg/dL) subjects. Over a 12 week test period, the probiotic group consumed 2g of powder daily containing dual probiotic strains, while the placebo group consumed the same without probiotics.

ELIGIBILITY:
Inclusion Criteria:

* nondiabetic (plasma fasting glucose, <126mg/dL; 2-hour plasma glucose, <200mg/dL)
* borderline to moderate hypertriglyceridemia (plasma triglyceride, 150-500 mg/dL)

Exclusion Criteria:

* lipid-lowering medications use
* any medications or supplement use
* any probiotics products use for the past 1 months
* dyslipidemia
* diabetes mellitus
* hypertension
* liver disease
* renal disease
* cardiovascular disease
* cerebrovascular disease
* pancreatitis
* cancer
* medication or alcohol abuse
* pregnant or breast feeding

Ages: 24 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
ApoA5-1131 genotype | at baseline
  ApoA5-1131 T>C

SECONDARY OUTCOMES:
Fasting glucose at baseline and 12-week follow-up | 12-week follow-up
  Serum fasting glucose (mg/dL)
Insulin at baseline and 12-week follow-up | 12-week follow-up
  Serum insulin (μIU/dL)
C-peptide at baseline and 12-week follow-up | 12-week follow-up
  Serum C-peptide (μEq/L)
Apolipoprotein A-V at baseline and 12-week follow-up | 12-week follow-up
  Plasma apolipoprotein A-V (ng/mL)
Triglyceride at baseline and 12-week follow-up | 12-week follow-up
  Serum triglyceride (mg/dL)
Free fatty acid at baseline and 12-week follow-up | 12-week follow-up
  Serum free fatty acid (μEq/L)

OTHER OUTCOMES:
LDL particle size at baseline and 12-week follow-up | 12-week follow-up
  Plasma LDL particle size (nm)
Serum high-sensitivity C-reactive protein at baseline and 12-week follow-up | 12-week follow-up
  Serum high-sensitivity C-reactive protein (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, PhD, Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Seoul, South Korea

REFERENCES:
- [Derived] Ahn HY, Kim M, Ahn YT, Sim JH, Choi ID, Lee SH, Lee JH. The triglyceride-lowering effect of supplementation with dual probiotic strains, Lactobacillus curvatus HY7601 and Lactobacillus plantarum KY1032: Reduction of fasting plasma lysophosphatidylcholines in nondiabetic and hypertriglyceridemic subjects. Nutr Metab Cardiovasc Dis. 2015 Aug;25(8):724-33. doi: 10.1016/j.numecd.2015.05.002. Epub 2015 May 14. PMID 26044516